CLINICAL TRIAL: NCT00208897
Title: Does Fluoxetine Reverse the Effects of Early Life Stress on the CNS Corticotropin-Releasing Factor System and Improve Psychological and Neuroendocrine Function?: A Therapy Outcome Study in Women With Childhood Abuse Experiences
Brief Title: Does Fluoxetine Have an Effect on the CNS CRF Systems in Women Abused in Childhood?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Dr. Christine Heim, Emory University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00001850; B1Y-MC-X176 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Early Life Stress; HPA-axis; CRF
MeSH Terms: conditions — Depressive Disorder, Major; Stress, Psychological | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
The primary objective of this project is to determine whether treatment with the SSRI, fluoxetine versus placebo reverses alterations in the central CRF system induced by early life stress experiences (i.e. childhood sexual and/or physical abuse) in cases with and without major depression. We also evaluate whether neuroendocrine changes after SSRI treatment correlate with clinical improvement.

DETAILED DESCRIPTION:
We compare indices of central CRF activity (i.e. ACTH and cortisol response to CRF stimulation test) before and after 8 weeks of treatment with either fluoxetine or placebo between women with a history of childhood abuse (early life stress, ELS) and current major depression (ELS/MDD), women with a history of childhood abuse without major depression (ELS/non-MDD), and women without a history of childhood abuse and major depression (non-ELS/MDD). Changes in neuroendocrine responses to CRF are correlated with psychological outcome measures. We hypothesize that treatment with fluoxetine will normalize altered neuroendocrine responsiveness in cases with ELS and that this normalization will be correlated with improvement of symptoms of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. For all subjects female gender;
2. For subjects assigned to the MDD groups, current DSM-IV diagnosis of MDD;
3. For subjects assigned to the early-life stress group, repeated (once per month or more for at least year) sexual or physical abuse before the age of 12 years by a perpetrator at least 5 years older at the time;
4. For all subjects, age of 18 to 45 years;
5. Regular menstrual cycle and assessment in the early follicular phase as verified by sex steroid measures.

Exclusion Criteria:

1. For all subjects, gender identity disorders;
2. For all subjects assigned to non-MDD groups, DSM-IV diagnosis of current MDD;
3. For all subjects assigned to the group without early-life stress, major stress experiences before the age of 12 years, such as separation from parents, neglect, parental loss, accidents, severe illness or natural disaster;
4. For all subjects, significant medical illness, such as gastrointestinal, neurological, endocrine, cardiovascular, pulmonary, renal, hepatic, immunological or hematological disease, organic brain disease, or cancer as determined by history, physical examination, ECG, and laboratory tests;
5. Pregnancy or nursing;
6. For all subjects, past or current presence of psychotic symptoms or bipolar disorder;
7. For all subjects, current presence of psychoactive substance abuse/dependency or eating disorders;
8. For all subjects, hormonal medication;
9. For all subjects, psychotropic medication in the four weeks prior to study entry;
10. For all subjects, inability to provide informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 1997-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Plasma ACTH and cortisol concentrations before and after administration of 1 microgram per kg ovine CRF | 6 hours

SECONDARY OUTCOMES:
Symptom Rating Scales for Depression, Anxiety and PTSD as well as general well-being | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Heim, PhD, Principal Investigator — Emory University-Dept. of Psychiatry and Behavioral Sciences
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia, United States